CLINICAL TRIAL: NCT02929654
Title: Assessment of Blood Glucose Monitoring Devices With New Insight Features
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 3150067
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Subject continue to use their own Blood Glucose Monitoring System ( BGMS) for 12 weeks.
  Interventions: Device: Subject's Own Blood Glucose Meter
- OneTouch Verio® (Experimental): Subjects use LifeScan provided BGMS (OneTouch Verio®) for 12 weeks
  Interventions: Device: OneTouch Verio®
- Intervention 02 (Experimental): Subjects use LifeScan provided BGMS (OneTouch Verio® Flex ) for 12 weeks.
  Interventions: Device: OneTouch Verio® Flex

INTERVENTIONS:
Device: OneTouch Verio® — Colour Enhanced Blood Glucose Meter.
  Arms: OneTouch Verio®
Device: OneTouch Verio® Flex — Colour Enhanced Blood Glucose Meter.
  Arms: Intervention 02
Device: Subject's Own Blood Glucose Meter — Subject's Own Blood Glucose Meter
  Arms: Control

SUMMARY:
To investigate whether novel insight features in new BGMs can improve glycemic control.

ELIGIBILITY:
Inclusion Criteria Summary:

* Diagnosed with T1DM or T2DM for ≥ 3 month prior to screening
* Currently performing SMBG at home for diabetes management decisions
* Willingness to notify the study staff if they become pregnant during the study
* Willing to sign an informed consent

Exclusion Criteria Summary:

* Is unlikely to be compliant with the diabetes regimen in the opinion of study staff
* Currently pregnant or planning pregnancy within duration of study or breast feeding; subjects who become pregnant during the study will be withdrawn
* Conflict of Interest

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
A1c change from baseline after 12 weeks | 12 weeks
  A1c change from baseline after 12 weeks in subjects using BGMs with color range indicator and/or pattern messaging tools (i.e., OneTouch Verio® Flex and OneTouch Verio® combined) compared to subjects with either T1 or T2DM using their current BGM, i.e., without color range indicator and/or pattern messaging tools.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Grady, Study Director — LifeScan Scotland
Locations (3):
- United Kingdom (3):
  - Diabetes Centre, Heartlands Hospital, Birmingham
  - NHS Lothian, Edinburgh
  - Highland Diabetes Institute, Inverness

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grady M, Katz LB, Levy BL. Use of Blood Glucose Meters Featuring Color Range Indicators Improves Glycemic Control in Patients With Diabetes in Comparison to Blood Glucose Meters Without Color (ACCENTS Study). J Diabetes Sci Technol. 2018 Nov;12(6):1211-1219. doi: 10.1177/1932296818775755. Epub 2018 May 31. PMID 29848106